CLINICAL TRIAL: NCT03148340
Title: VITAL: Volumetric Integral Phase-shift Spectroscopy (VIPS) for the Noninvasive Detection of Hemispheric Bioimpedance Asymmetry in Acute Brain Pathology
Brief Title: Volumetric Integral Phase-shift Spectroscopy for Noninvasive Detection of Hemispheric Bioimpedance Asymmetry in Acute Brain Pathology
Acronym: VITAL
Status: Completed | Type: Observational
Sponsor: Cerebrotech Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CH006
Record Dates: First submitted 2017-05-08; First posted 2017-05-11 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Stroke; Stroke, Acute; Ischemic Stroke; Hemorrhage; Clot (Blood); Brain; Subarachnoid Hemorrhage; Cerebral Infarction; Cerebral Hemorrhage; Cerebral Stroke; Intracerebral Hemorrhage; Intracerebral Injury
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhage; Intracranial Thrombosis; Subarachnoid Hemorrhage; Cerebral Infarction; Cerebral Hemorrhage; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VIPS monitoring group: The study population will consist of adult patients presenting for evaluation of acute brain pathology,
  Interventions: Diagnostic Test: VIPS Monitoring

INTERVENTIONS:
Diagnostic Test: VIPS Monitoring — Bioimpedance asymmetry
  Other Names: CMS

SUMMARY:
The purpose of this study is to assess the ability of the Fluids Monitor to detect hemispheric bioimpedance asymmetry associated with acute brain pathology in patients presenting with suspected Acute Ischemic Stroke (AIS).

DETAILED DESCRIPTION:
A prospective non-significant-risk (NSR) multi-site observational study. This study will examine up to 318 subjects undergoing evaluation for acute brain pathology who directly arrive at, or are transferred to, the participating sites.

ELIGIBILITY:
Inclusion Criteria:

1. Must be at least 18 years of age.
2. Being evaluated for acute ischemic stroke.
3. Able to safely wear the study device for up to 2 minutes per reading.
4. Have NIHSS performed before before study device monitoring.
5. Must be able to provide written Informed Consent (either self or via an LAR) at any point during the hospital stay, or if unable to provide such consent, must have permission granted by the governing IRB to enroll in the study (i.e., waiver of consent).

Exclusion Criteria:

1. Known or suspected traumatic brain injury, either closed or penetrating.
2. Contraindication to neuroimaging, such as a contrast allergy, or other condition that prohibits CT, MRI, and/or angiography.
3. Presence of any implanted electro-stimulating devices in the head and neck.
4. Presence of any large metallic craniofacial implants, such as bone fixation plates, mesh, et cetera. (Note that small metallic objects, such an aneurysm coils, are acceptable.)
5. Presence of an intracranial pressure monitor or any other similar sensor that may compromise the placement of the investigational device.
6. Under arrest or otherwise in custody.
7. Inability to wear the investigational device (skin lesions on scalp, previous intracranial surgeries, etc.).
8. Pregnant or nursing.
9. Any other condition, which in the judgment of the PI would prevent the patient from completing the study or tolerating monitoring sessions and brain imaging, such as mental illness, severe agitation, or hemodynamic instability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females, aged 18 years or older, who are undergoing evaluation for acute ischemic stroke
Sampling Method: Non-Probability Sample
Enrollment: 287 (Actual)
Dates: Start 2017-04-14 (Actual); Primary Completion 2018-05-10 (Actual); Study Completion 2018-07-15 (Actual)

PRIMARY OUTCOMES:
Hemispheric bioimpedance asymmetry detection | At the time of VIPS monitoring - day 0
  The primary outcome will be the device's ability to detect hemispheric bioimpedance asymmetry associated with acute brain pathology in a population of patients presenting with symptoms consistent with AIS

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Lyerly Baptist, Inc, Jacksonville, Florida
  - University of Buffalo, Buffalo, New York
  - The Mount Sinai Hospital, New York, New York
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee Health Science Center, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith WS, Lev MH, English JD, Camargo EC, Chou M, Johnston SC, Gonzalez G, Schaefer PW, Dillon WP, Koroshetz WJ, Furie KL. Significance of large vessel intracranial occlusion causing acute ischemic stroke and TIA. Stroke. 2009 Dec;40(12):3834-40. doi: 10.1161/STROKEAHA.109.561787. Epub 2009 Oct 15. PMID 19834014
- [Background] Nogueira RG, Zaidat OO, Castonguay AC, Haussen DC, Martin CO, Holloway WE, Mueller-Kronast N, English J, Linfante I, Dabus G, Malisch TW, Marden FA, Bozorgchami H, Xavier A, Rai AT, Froehler MT, Badruddin A, Nguyen TN, Taqi MA, Abraham MG, Janardhan V, Yoo AJ, Shaltoni H, Abou-Chebl A, Chen PR, Britz GW, Novakovic R, Nanda A, Kaushal R, Issa MA, Frankel MR, Gupta R. Rescue Thrombectomy in Large Vessel Occlusion Strokes Leads to Better Outcomes than Intravenous Thrombolysis Alone: A 'Real World' Applicability of the Recent Trials. Interv Neurol. 2016 Sep;5(3-4):101-110. doi: 10.1159/000445809. Epub 2016 May 27. PMID 27781037
- [Background] Goyal M, Menon BK, van Zwam WH, Dippel DW, Mitchell PJ, Demchuk AM, Davalos A, Majoie CB, van der Lugt A, de Miquel MA, Donnan GA, Roos YB, Bonafe A, Jahan R, Diener HC, van den Berg LA, Levy EI, Berkhemer OA, Pereira VM, Rempel J, Millan M, Davis SM, Roy D, Thornton J, Roman LS, Ribo M, Beumer D, Stouch B, Brown S, Campbell BC, van Oostenbrugge RJ, Saver JL, Hill MD, Jovin TG; HERMES collaborators. Endovascular thrombectomy after large-vessel ischaemic stroke: a meta-analysis of individual patient data from five randomised trials. Lancet. 2016 Apr 23;387(10029):1723-31. doi: 10.1016/S0140-6736(16)00163-X. Epub 2016 Feb 18. PMID 26898852
- [Background] Saver JL, Goyal M, van der Lugt A, Menon BK, Majoie CB, Dippel DW, Campbell BC, Nogueira RG, Demchuk AM, Tomasello A, Cardona P, Devlin TG, Frei DF, du Mesnil de Rochemont R, Berkhemer OA, Jovin TG, Siddiqui AH, van Zwam WH, Davis SM, Castano C, Sapkota BL, Fransen PS, Molina C, van Oostenbrugge RJ, Chamorro A, Lingsma H, Silver FL, Donnan GA, Shuaib A, Brown S, Stouch B, Mitchell PJ, Davalos A, Roos YB, Hill MD; HERMES Collaborators. Time to Treatment With Endovascular Thrombectomy and Outcomes From Ischemic Stroke: A Meta-analysis. JAMA. 2016 Sep 27;316(12):1279-88. doi: 10.1001/jama.2016.13647. PMID 27673305
- [Background] Kodankandath TV, Wright P, Power PM, De Geronimo M, Libman RB, Kwiatkowski T, Katz JM. Improving Transfer Times for Acute Ischemic Stroke Patients to a Comprehensive Stroke Center. J Stroke Cerebrovasc Dis. 2017 Jan;26(1):192-195. doi: 10.1016/j.jstrokecerebrovasdis.2016.09.008. Epub 2016 Oct 12. PMID 27743926
- [Background] Jauch EC, Saver JL, Adams HP Jr, Bruno A, Connors JJ, Demaerschalk BM, Khatri P, McMullan PW Jr, Qureshi AI, Rosenfield K, Scott PA, Summers DR, Wang DZ, Wintermark M, Yonas H; American Heart Association Stroke Council; Council on Cardiovascular Nursing; Council on Peripheral Vascular Disease; Council on Clinical Cardiology. Guidelines for the early management of patients with acute ischemic stroke: a guideline for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2013 Mar;44(3):870-947. doi: 10.1161/STR.0b013e318284056a. Epub 2013 Jan 31. PMID 23370205
- [Background] Hastrup S, Damgaard D, Johnsen SP, Andersen G. Prehospital Acute Stroke Severity Scale to Predict Large Artery Occlusion: Design and Comparison With Other Scales. Stroke. 2016 Jul;47(7):1772-6. doi: 10.1161/STROKEAHA.115.012482. Epub 2016 Jun 7. PMID 27272487
- [Background] John S, Stock S, Masaryk T, Bauer A, Cerejo R, Uchino K, Winners S, Rasmussen P, Hussain MS. Performance of CT Angiography on a Mobile Stroke Treatment Unit: Implications for Triage. J Neuroimaging. 2016 Jul;26(4):391-4. doi: 10.1111/jon.12346. Epub 2016 Mar 30. PMID 27028362
- [Background] Rojas R, Rubinsky B, Gonzalez CA. The effect of brain hematoma location on volumetric inductive phase shift spectroscopy of the brain with circular and magnetron sensor coils: a numerical simulation study. Physiol Meas. 2008 Jun;29(6):S255-66. doi: 10.1088/0967-3334/29/6/S22. Epub 2008 Jun 11. PMID 18544824
- [Background] Zuckerman SL, Sivaganesan A, Zhang C, Dewan MC, Morone PJ, Ganesh Kumar N, Mocco J. Maximizing efficiency and diagnostic accuracy triage of acute stroke patients: A case-control study. Interv Neuroradiol. 2016 Jun;22(3):304-9. doi: 10.1177/1591019915622167. Epub 2016 Feb 2. PMID 26842606